CLINICAL TRIAL: NCT00908986
Title: Open Label Pilot Trial of Rituximab in Lupus Membranous Nephritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: Northwell Health (Other)
Responsible Party: Cynthia Aranow, MD, Feinstein Institute for Medical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U2971g
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Lupus Nephritis
Keywords: Lupus Membranous Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): Subjects receive rituximab in an open label manner
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 q week x 4; repeated in 6 months
  Other Names: Rituxan

SUMMARY:
The objective of this study is to assess the as efficacy of rituximab as induction therapy in membranous lupus nephritis. Safety and tolerability will additionally be assessed. Subjects will receive open-label 2 courses of rituximab at baseline and at 6 months. They will be followed monthly for 18 months to assess response and durability of response.

The hypothesis: B cell depletion will be an effective safe and well tolerated treatment for membranous lupus nephritis (Class V).

ELIGIBILITY:
Inclusion Criteria:

* Age of a minimum of 18 years old
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Negative serum pregnancy test (for women of child bearing potential)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* Diagnosis of SLE per current ACR classification criteria (at least 4 of 11 criteria)
* Base line proteinuria >2g/24h
* Kidney biopsy within 12 months of enrollment with membranous L.N. (ISN/RPS V)
* Full dose ACE inhibition (or ARB) for a minimum of 8 weeks at day 0. Patients may be on less than full dose due to lack of tolerability
* Stable < 0.5mg/kg corticosteroid dose in the 4 weeks prior to screening (including no corticosteroid)
* Background immunosuppressives to include azathioprine, cyclosporine A, mycophenolate mofetil, methotrexate and/or an anti-malarial for > 6 months with stable dose(s) for 1 month prior to screening/enrollment will be allowed. Patients receiving cyclophosphamide and/or leflunomide will be excluded from this study.

Exclusion Criteria:

* Treatment with cyclophosphamide within 3 months of screening
* Use of high dose steroids (>0.5 mg/kg/ day) in the 4 weeks prior to screening
* ANC < 1.5 x 103
* Hemoglobin: < 8.0 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* Positive Hepatitis B or C serology (Hep B Surface antigen and Hep C antibody)
* History of positive HIV (HIV conducted during screening if applicable)
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* Previous treatment with Natalizumab (Tysabri®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids (>0.5 mg/kg/ day ) or unstable steroid dose in the past 4 weeks
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
* Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Efficacy at 6 months post treatment and durability of response at 12 months post treatment will be determined by: reduction in 24 hour urinary protein excretion, reciprocal creatinine, urinary sediment | 12 months

SECONDARY OUTCOMES:
Change from baseline at 6 and 12 months in non-renal SLE disease activity (BILAG), lupus serologies (anti-dsDNA antibodies) and complement consumption (C3, C4), serum albumin, cholesterol, triglycerides | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Principal Investigator — Feinstein Institute for Medical Research